CLINICAL TRIAL: NCT05230563
Title: A Clinical Study of LUNG-CT CAD Decision Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TaiHao Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TaiHao LUNG-CTCAD CCH 210129
Record Dates: First submitted 2022-01-14; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participating clinicians will perform lung nodule detection on 200 cases of lung low-dose computed tomography images
- Experimental Group - with the aid of "Taihao" lung CT decision support system (Experimental): Participating clinicians will perform lung nodule detection on 200 cases of lung low-dose computed tomography images with the aid of "Taihao" lung CT decision support system
  Interventions: Device: Ti-LUNG

INTERVENTIONS:
Device: Ti-LUNG — Participating clinicians will perform two image interpretations on all cases. One period the clinicians only will perform lung nodule detection on chest CT images, and the other period will perform lung nodule detection on chest CT images with the aid of "Taihao" lung CT decision support system. In each interpretation, all lung nodule is marked by each radiologist. This test collects chest computerized tomography cases for computer analysis, and evaluates whether the "TaiHao" lung CT decision support system helps doctors make more accurate diagnoses.
  Arms: Experimental Group - with the aid of "Taihao" lung CT decision support system

SUMMARY:
This product is a computer-aided detection software designed to assist clinicians in detecting lung nodules in chest computer tomography. This product receives from PACS, radiology information system or directly from computer tomography scanner. After receiving the image, the product performs image analysis and provides a mark of suspected lung nodules. Users can use existing medical image capture and transmission systems or reading software to view these annotations on the workstation.

The main purpose of this trial is to verify that when clinicians perform chest CT pulmonary nodule detection, compared to only diagnosis based on chest CT images, whether the "Taihao" lung CT decision support system helps to improve the diagnostic efficiency of clinicians.

The secondary purpose is to evaluate that when clinicians perform chest CT pulmonary nodule detection, compared to only diagnosis based on chest CT images, whether the "Taihao" lung CT decision support system helps to improve the sensitivity, specificity, and image interpretation time (Reading Time) of clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Cases of men or women aged between 20 and 89.
* At Changhua Christian Hospital or Yuanlin Christian Hospital, expert (qualified for interpretation of chest computed tomography lung nodules) confirms that the original low-dose computed tomography image had pulmonary nodules (part solid nodule, solid nodule, and pulmonary nodules greater than or equal to 3 mm), and verified that it is as a true nodule through follow-up clinical imaging examination or clinical determination, or
* At Changhua Christian Hospital or Yuanlin Christian Hospital, the subject has undergone a low-dose lung computed tomography and a physician (qualified for interpretation of chest computed tomography lung nodules) confirmed that there are no lung nodules on the computed tomography scan.

Exclusion Criteria:

* The computerized tomography of the lungs and obvious administrative or technical errors.
* A physician (qualified for interpretation of chest CT pulmonary nodules) confirms cases with severe infections such as tuberculosis and pneumonia from source report or other medical records.
* A physician (qualified for interpretation of chest CT pulmonary nodules) confirms cases with lung fibrosis such as pneumoconiosis from source report or other medical records.
* Test cases used when training physicians to use the lung computer tomography decision support system.

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC Curve(AUC) | 4 months
  The primary outcome measure is the area under the receiver operating characteristic (ROC) curve of the radiologists, also known as c statistic.

SECONDARY OUTCOMES:
Sensitivity | 4 months
  True Positive / True Positive + False Negative
Specificity | 4 months
  True Negative / False Positive + True Negative
Interpretation time | 4 months
  Reading Time of clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tai Chen, Ph.D, Principal Investigator — Study Director
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua County, Taiwan